CLINICAL TRIAL: NCT06133790
Title: Assessment of Genomic Alterations and Profiles of Expression in HPV+ Versus HPV Head and Neck Cancers
Brief Title: Profiles of Expression in HPV+ Versus HPV Head and Neck Cancers
Acronym: HPVNGS
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00936-39
Record Dates: First submitted 2023-10-23; First posted 2023-11-15 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA is extracted from biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HPV + Group: Patients with positive HPV diagnosis
  Interventions: Genetic: PCR - Immunohistochemistry - Immunolabelling
- HPV - Group: Patients with negative HPV diagnosis
  Interventions: Genetic: PCR - Immunohistochemistry - Immunolabelling

INTERVENTIONS:
Genetic: PCR - Immunohistochemistry - Immunolabelling — Genetic analysis will be conducted on biopsy to define molecular profile of head and neck tumors

SUMMARY:
Squamous cell cancers of the head and neck are classically correlated to excessive consumption of alcohol and tobacco and have a rather poor prognosis. However, the incidence of Head and Neck cancers in patients without alcohol-smoking risk factor has continued to increase in recent years, in relation to more and more frequent HPV contamination.

Some studies show a difference in the expression of certain genes within the two groups of tumors (HPV+ and HPV-) including some that confer sensitivity to certain chemotherapies and others to radiotherapy. However, patients with HPV+ Head and Neck cancers are treated according to the same referential as HPV- Head and Neck cancers. There is therefore a real need for studies identifying predictive markers in order to be able to offer patients a more effective suitable and less invasive treatment.

DETAILED DESCRIPTION:
Head and neck cancers are the sixth most common cancer common worldwide causing more than 380,000 deaths each year. More than 90% of these cancers are carcinomas epidermoids arising from the mucosal surfaces of the cavity oral cavity, oropharynx and larynx.

Squamous cell cancers of the head and neck are classically correlated with risk factors linked to excessive consumption of alcohol and tobacco and have a rather poor prognosis (mainly HPV (Human Papilloma Virus) negative patients).

However, the incidence of Head and Neck cancers in patients without alcohol-smoking risk factor has continued to increase in recent years, in relation to more and more frequent HPV contamination. Evolution of oral sexual practices seems to be one of the explanations for the progression of these cases of oropharyngeal squamous cell carcinoma and oral cavity HPV positive.

Some studies show a difference in the expression of certain genes within the two groups of tumors (HPV+ and HPV-) including some that confer sensitivity to certain chemotherapies (CCND1, TYMS) and others to radiotherapy (RBBP4). However, patients with HPV+ Head and Neck cancers are treated according to the same referential as HPV- Head and Neck cancers. There is therefore a real need for studies identifying predictive markers in order to be able to offer patients a more effective suitable and less invasive treatment. This is the context of this research project.

ELIGIBILITY:
Inclusion Criteria:

* Patient with oropharyngeal squamous cell carcinoma or the oral cavity histologically proven.
* Primary tumor for which a biopsy or excision is required available and sufficient to carry out molecular analysis

Exclusion Criteria:

- Patient with Head and Neck cancer other than oropharyngeal or oral cavity squamous cells carcinomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Head and Neck cancer and HPV diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Molecular profile of oropharyngeal or oral cavity HPV positive and negative tumors | 1 day
  Molecular profile of tumors will be established with analysis of 87 "Hotspot" genes, full length analysis of 48 genes, copy number analysis of 43 genes and gene fusion (inter and intra genic) of 51 genes.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme PARIS, MD, Principal Investigator — Hôpital privé de Clairval
Locations (1):
- Hôpital Privé Clairval, Marseille, France

IPD SHARING:
Plan to Share IPD: No